CLINICAL TRIAL: NCT06871514
Title: 2-DECIDE: A Stepped-Wedge Multicenter Study on the Effectiveness of a Multicomponent Intervention With Shared Decision-Making to Improve Cardiovascular Risk Management in Adults With Established Atherosclerotic Cardiovascular Disease
Brief Title: Effectiveness of Decision Support for Cardiovascular Risk Management in People With Cardiovascular Disease
Acronym: 2-DECIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: dr.Frank L.J. Visseren (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, dr.Frank L.J. Visseren, Prof. dr. F.L.J. Visseren, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24U-1636
Record Dates: First submitted 2025-02-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerotic Cardiovascular Diseases; Shared-decision Making

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Clinical Trial: All centers will start with care as usual. At randomized intervals, they will switch to application of the 2-DECIDE intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other)
  Interventions: Other: No Intervention: usual care
- 2-DECIDE intervention (Experimental)
  Interventions: Other: 2-DECIDE intervention: decision support for cardiovascular risk management

INTERVENTIONS:
Other: 2-DECIDE intervention: decision support for cardiovascular risk management — The 2-DECIDE intervention consists of:
  * Training of healthcare providers in implementing shared decision-making during clinical consultations.
  * At least one initial extended outpatient consultation with a trained physician to ensure adequate time for actual understanding of treatment options.
  * Decision support based on U-prevent
  * Clear communication to the patient is provided in an easily comprehensible format, including pre-visit information, and a post-visit handout of the information and decisions made using the U-prevent medical device. Additionally, the general practitioner receives a letter detailing the outcome and rationale of the shared decision, along with the individual estimates that have informed the treatment choice.
  Arms: 2-DECIDE intervention
Other: No Intervention: usual care — Usual care
  Arms: Usual care

SUMMARY:
This study aims to improve the way patients with cardiovascular diseases are informed about their treatment options. It explores methods to support shared decision-making between patients and doctors. In some cases, doctors will take extra time to discuss treatment options in detail. To assess the impact, some patients will be asked to complete questionnaires after their clinic visits.

ELIGIBILITY:
Inclusion criteria:

* Established ASCVD

  * At least 30 days since last CVD event and/or the diagnosis of ASCVD. If no CVD events have occurred, imaging confirming ASCVD must have been conducted at least 30 days prior.
  * Documented ASCVD (defined according to the 2021 European Society of Cardiology guideline), which includes ASCVD established clinically or demonstrated unequivocally by imaging:
* Clinically documented ASCVD includes previous myocardial infarction, acute coronary syndrome, coronary revascularization (Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Surgery (CABG)), and other arterial revascularization procedures, ischemic stroke or transient ischemic attack, and peripheral artery disease (from Fontaine stage II). Angina pectoris (stable) without imaging evidence of atherosclerosis does not qualify as ASCVD.
* ASCVD unambiguously identified through imaging, includes significant stenosis (>50%) on coronary angiography, computed tomography angiography, or carotic ultrasound. It also includes aortic aneurysms measuring ≥3cm. Only Carotid Intima-Media Thickness measurements (cIMT), Coronary Artery Calcium scoring or abnormal ankle-brachial index scores without evidence of stenosis, do not qualify as ASCVD.
* Age 40-80 years (to allow for individual risk predictions with the SMART2 model
* Patient attending the Cardiology or Vascular Medicine outpatient clinic
* Sufficient understanding of the Dutch language (due to the questionnaires being administered in Dutch).
* Written informed consent must be provided. Although the proposed intervention is not subject to the WMO, informed consent is required for the collection and processing of data, including the distribution of questionnaires.

Exclusion criteria:

* Patients currently participating in other interventional medication studies, or studies that directly affect the therapy plan
* Remaining life expectancy of less than 2 years as assessed by a consulting healthcare professional (these patients have no indication for cardiovascular risk management)
* Patients for whom individual risk predictions with the SMART2 model are not feasible:

  * Systolic Blood Pressure (SBP) <90 mmHg or >200 mmHg
  * Total cholesterol <2.5mmol/L or >8 mmol/L
  * High-Density Lipoprotein (HDL) cholesterol <0.6mmol/L or >2.5 mmol/L
  * Low-Density Lipoprotein (LDL) <0.1 mmol/L or >7.4 mmol /L
  * Estimated Glomerular Filtration Rate (eGFR) <30ml/min/1.73m2 or dialysis
  * Active treatment for malignity, pregnancy, history of organ transplantation, or liver failure
* Previous participation in 2-DECIDE

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
10-year residual cardiovascular disease risk | At 12 months from enrollment
  Calculated using the SMART2 risk model
Adherence to medication | At 12 months from enrollment
  Assessed using data on medication dispensing data via Stichting Farmacotherapeutische Kengetallen (SFK) linkage, which connects individual pharmacy records across the Netherlands
Beliefs underlying adherence | Baseline and at 12 months from enrollment
  Assessed using the Beliefs about Medicines Questionnaire (BMQ), consisting of BMQ-General (8 items) and BMQ-Specific (11 items). Items are rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Subscale scores are summed, and difference scores between subscales are calculated. In BMQ-Specific, a positive score indicates perceived benefits outweigh concerns about medicination. In BMQ-General, a positive score indicates trust in medication and prescribing outweighs negative perceptions of medicines in general.
Knowledge and motivation in patient | Baseline and at 12 months from enrollment
  Assessed using the Patient Activation Measure ® (PAM-13 ®), an empirical interval scale from 0 to 100, corresponding to four patient activation levels. Levels 1-2 indicate lower activation, while Levels 3-4 indicate higher activation.
Experienced shared-decision making | At baseline (0 months from enrollment)
  Assessed using the 9-item Shared Decision Making Questionnaire (SDM-Q9), rated on a 6-point scale (0 = completely disagree, 5 = completely agree). The total raw score (0-45) is transformed to a 0-100 scale, with higher scores indicating greater experienced shared decision-making by the patient
Decisional conflict | At baseline (0 months from enrollment)
  Assessed using the 16-item Decisional Conflict Scale (DCS), rated on a 5-point scale (0 = strongly agree, 4 = strongly disagree). Scores are transformed to a 0-100 scale, where higher scores indicate greater decisional conflict.
Quality of life (as measured with PROMIS) | At 12 months from enrollment
  Assessed using two shorts form of the Patient-Reported Outcomes Measurement Information System (PROMIS): Global Health Form and Physical Function. Scores are standardized T-scores (mean = 50, SD = 10), with higher scores indicating better physical function and overall health.

SECONDARY OUTCOMES:
Consultation efficiency (healthcare providers' perceived acceptability, appropriateness, and feasibility of the intervention) | Within 1 month of last inclusion of consulting healthcare provider
  Measured using the Acceptability of Intervention Measure, Intervention Appropriateness Measure, & Feasibility of Intervention Measure. Each measure consists of four items rated on a 5-point Likert scale (1 = Completely disagree, 5 = Completely agree). Scores are averaged (range: 1-5), with higher scores indicating greater acceptability, appropriateness, and feasibility. These measures will be completed once by the consulting healthcare providers at the end of the inclusion period of the intervention phase.
Cost-effectiveness composite | Short-term costs observed through the iMCQ/iPCQ questionnaire (administered at 3, 6, and 12 months) will be used to model long-term costs and benefits, projected over a lifetime horizon.
  Modelled long-term cost and benefit outcomes. In line with the Dutch recommendations for performing cost-effectiveness analyses, a lifetime horizon will be used (a modelled approach, based on extrapolation of short-term observed costs). This modelling will be performed using study-specific data, supplemented with Dutch data on event and care costs across this population for a more stable estimate (UCC-SMART cohort linked to VEKTIS cost data)
Prescription rates of cardiovascular disease preventive treatments | At 12 months from enrollment
Healthcare costs | From baseline to the end of follow-up at 12 months. (the questionnaire is administered at 3, 6 and 12 months from enrollment)
  Medication and healthcare consumption, using an adjusted version of the iMTA Medical Consumption Questionnaire (iMCQ) and iPCQ (Productivity Cost Questionnaire)
Quality of life (to inform cost-effectiveness analyses) | At 12 months from enrollment
  Assessed using EuroQol (EQ-5D-5L), to inform cost-effectiveness analyses. The EQ-5D-5L measures health across five dimensions, each with five levels of perceived problems. A summary index is calculated by applying weights to each level and deducting them from 1 (full health), with higher scores indicating better health. Index values support economic evaluations of healthcare interventions.

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Radboudumc, Nijmegen
  - HagaZiekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No